CLINICAL TRIAL: NCT00849745
Title: Nonmyeloablative Allogeneic Peripheral Blood Stem Cell Transplantation for Severe Autoimmune Diseases
Brief Title: Nonmyeloablative Allo Stem Cell Transplant for Severe Autoimmune Diseases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010324
Record Dates: First submitted 2009-02-22; First posted 2009-02-24 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Systemic Lupus Erythematosus; Systemic Sclerosis
Keywords: severe autoimmune diseases; allogeneic stem cell transplant
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Autoimmune Diseases | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Systemic Lupus Erythematosus (Experimental): Nonmyeloablative allogeneic stem cell transplant
  Patients must:
  * Satisfy the American College of Rheumatology (ACR) criteria for the diagnosis of SLE
  * Have Lupus nephritis, refractory and severe seizures or encephalopathy, severe pulmonary involvement, transfusion-dependent cytopenias, catastrophic antiphospholipid syndrome or vasculitis and/or immune complex deposition causing end-organ signs or symptoms.
  * Have received a trial of corticosteroids equivalent to prednisone greater than or equal to 0.5 mg/kg/d for at least one month
  * Have received a trial of IV cyclophosphamide pulse greater than 500 mg/square meter at least once within the previous 6 months, unless contraindicated because of severe cytopenias or intolerance.
  Interventions: Procedure: Nonmyeloablative allogeneic stem cell transplant
- Systemic Sclerosis (Experimental): Nonmyeloablative allogeneic stem cell transplant
  Patients must:
  * Have diagnosis of SSc as defined by American College of Rheumatology and at high-risk for fatal outcome.
  * Have (1) both a and b below and (2) at least one of c, d, or e.
  * Diffuse cutaneous scleroderma with skin score of >= 16
  * Duration of systemic sclerosis <= 3 years from the onset of first non-Raynaud's symptom.
  * Presence of interstitial or pulmonary vascular lung involvement (FVC or DLCO <70% of predicted) especially with evidence of alveolitis (abnormal bronchoalveolar lavage or high-resolution chest CT scan).
  * Presence of myocardial disease
  * History or presence of proteinuria > 500 mg/24 hrs or serum creatinine > the upper limit of normal.
  Interventions: Procedure: Nonmyeloablative allogeneic stem cell transplant

INTERVENTIONS:
Procedure: Nonmyeloablative allogeneic stem cell transplant — Prior to receiving Campath-1H, patients will be premedicated with Benadryl 50 mg IV or PO, and acetaminophen 650 mg orally. Hydrocortisone 100 mg IV is given on the first day of Campath. The preparative regimen will begin on day -5 and consist of 4 days of daily fludarabine at 30 mg/m2/d infused over 30 minutes, cyclophosphamide 500 mg/m2/d infused over 1 hour, 5 days of Campath-1H at 20 mg/d in 250 ml of D5 normal saline or normal saline infused over 3 hours. The mixed dosage of chemotherapy may be rounded off to within +/- 5% of the calculated dose, and doses of fludarabine and cyclophosphamide will be based on adjusted ideal body weight. IV hydration and diuretics will be used to maintain adequate urine output during and after administration of cyclophosphamide.
  Other Names: Campath-1H

SUMMARY:
Autoimmune diseases present a special challenge to clinicians and the aim of this protocol is to serve as a last-line effort for patients with unmanageable disease. The primary purpose of this study is to assess feasibility in terms of toxicity and engraftment of a less toxic, nonablative conditioning regimen of Campath-1H, moderate dose fludarabine, and cyclophosphamide for patients with severe autoimmune diseases.

DETAILED DESCRIPTION:
Our targeted illnesses are:

* Systemic lupus erythematosus (SLE): SLE can involve virtually any organ system, but most commonly involves various combinations of arthritis, dermatitis, glomerulonephritis, central nervous system manifestations and hematologic complications. Although the overall five and ten-year survival rates in SLE are 86% and 80%, respectively, these rates are reduced to 60% and 50%, respectively, in patients with poor prognosis SLE (proliferative glomerulonephritis with chronic changes, elevated serum creatinine, nephrotic syndrome, anemia, low serum C3, inadequate response to treatment).
* Systemic sclerosis (SSc): SSc is a condition divided into two forms (diffuse and limited) characterized by excessive and often relentless fibrosis in skin and internal organs. Visceral involvement can manifest as esophageal hypomotility, interstitial lung disease, pulmonary hypertension and renal failure. There is no satisfactory treatment for systemic sclerosis (SSc), which in its diffuse form has a 5-year mortality of 40%, similar to many malignancies. In clinical trials, alpha-interferon did not demonstrate a clinically significant effect and low dose methotrexate showed conflicting results.

ELIGIBILITY:
Patient Inclusion Criteria:

* Performance status must be CALGB PS 0, 1, or 2 (or Karnofsky 40-100%)
* Patients must have a 6/6 HLA-matched related donor who is evaluated and deemed able to provide PBSCs and/or marrow by the transplant team.
* Patients must meet the following laboratory parameters (unless due to disease status as determined by the treating physician):

  * Hepatitis A, B and C status will be tested prior to therapy, but results will not exclude patients from participation (if positive, patients will be told they are at higher risk of adverse effects from allogeneic transplantation).
  * Bilirubin less than 6 times the upper limit of normal
  * Liver transaminases (AST, ALT) and alkaline phosphatase less than 10 times the upper limit of normal (unless due to active myositis)
  * Patients with a creatinine greater than 2.5 times the upper limit of normal are eligible, but will be told that they are at greater risk for kidney damage that could possibly result in temporary or even permanent dialysis.
* Patients of childbearing potential must agree to use some form of adequate birth control during the periods they receive chemotherapy and any post-chemotherapy medications related to the transplant. Females of child bearing potential must have a negative serum B-HCG within 1 week of starting therapy.
* Patients between the ages of 18 and 69, inclusive are eligible for this trial.
* Patients must also have a resting MUGA (preferred) or ECHO and PFTs with DLCO performed before transplant and found to be acceptable according to the treating institution's guidelines. Recommended minimum standards include an EF greater than 35% and corrected DLCO greater than 35% for this less toxic regimen. If lower than this, single patient exemption may be sought.
* Patients must have both a disease-specialist (rheumatologist/immunologist, or neurologist) physician and a bone marrow transplant physician evaluation at the treating center before a patient is considered eligible. Both specialists must agree that the patient is a candidate for transplantation and patients with SLE must have failed standard therapies.

Exclusion Criteria:

* Pregnant or lactating women
* Active uncontrolled infection
* Patients who are serologically true-positive for HIV
* Patients with other major medical or psychiatric illnesses, which the treating physician feels, could seriously compromise tolerance to this protocol
* Uncontrolled hypertension (BP > 100 diastolic despite treatment with maximum doses of at least 3 simultaneous or concurrent antihypertensives over a 2-month period)
* Uncontrolled malignant arrythmias or clinical evidence of congestive heart failure (New York Class IV)

6/6 HLA-Matched Related PBSC Donor Inclusion/Exclusion Criteria:

* Adult donors must be capable of providing informed consent; Potential donors under the age of 18 must have a 'single patient exemption' approved by the IRB and the donor and a guardian must provide assent.
* Donor must be 6/6 HLA matched, and related to the patient.
* Donor must not have any medical condition which would make apheresis and G-CSF administration more than a minimal risk, and should have the following:

  1. Adequate cardiac function by history and physical examination. Those with a history of cardiac problems should undergo a stress evaluation or be evaluated by a cardiologist and deemed eligible to donate.
  2. bilirubin and hepatic transaminases < or equal to 2.5 x ULN,
  3. adequate hematologic parameters including a hematocrit > 35% for males and 33% for females, white blood cell count of > or equal to 3,000, and platelets > or equal to 80,000.
  4. Donors with a known allergy to E. coli-derived products are ineligible for mobilization with G-CSF.
* Females of childbearing potential should have a negative serum beta-HCG test within 1 week of beginning G-CSF.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Engraftment | 24 months
Graft versus Host Disease | 45 days
Toxicity | 45 days
  Occurrence of Grade 3-4 adverse events
Mortality | 24 months
  Occurrence of deaths

SECONDARY OUTCOMES:
Response Rate | 24 months
Immune Function Post-engraftment | 24 months
Progression Free Survival | 24 months
Overall Survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Keith Sullivan, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States